CLINICAL TRIAL: NCT06939946
Title: Early Feasibility Study on Intraoperative Parathyroid Gland (PTG) Identification Using a Hand-Held Imager (HHI)
Brief Title: Intraoperative Parathyroid Gland (PTG) Identification Using a Hand-Held Imager (HHI)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The NIH-funded project period has come to an end.
Sponsor: OPTOSURGICAL, LLC (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00224302
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Disease; Thyroid Surgery; Parathyroid Gland
Keywords: Thyroid surgery; Parathyroid fluorescence; Indocyanine Green
MeSH Terms: conditions — Thyroid Diseases | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Parathyroid auto-florescence imaging (Experimental): Patients undergoing open thyroid surgery
  Interventions: Device: Parathyroid auto-fluorescence imaging; Drug: Indocyanine green

INTERVENTIONS:
Device: Parathyroid auto-fluorescence imaging — All enrolled patients for thyroid surgery, once the thyroid gland is removed the device will be used to identify the parathyroid glands.
  Other Names: hANDY-i; Hand-Held Imager
Drug: Indocyanine green — For a select group of patients when deemed necessary by the surgeon, and when one or more parathyroid gland appear to be de vascularized ICG will be administered, A dosage of 5 mg will be injected into a peripheral IV line, followed by fluorescence imaging to determine the perfusion status of the gland.
  Other Names: ICG

SUMMARY:
It is often challenging to tell apart the parathyroid glands from the surrounding area such as lymph nodes, fat and thyroid tissue. If the surgeons are not able to tell where the parathyroid glands are, they might accidentally be removed or damaged. This can lead to complications such as hypocalcemia (low calcium level) requiring treatment and sometimes lead to longer hospital stay. This study is designed to test a new method (a non-invasive hand-held imaging device) to assist surgeons in identifying the parathyroid glands, in order to decrease the rate of post-operative complication.

DETAILED DESCRIPTION:
In thyroid surgeries, it is often difficult to visually distinguish parathyroid glands (PTGs) from the surrounding anatomical structures in surgeries because of their small size and appearance that is similar to lymph nodes, fat, and thyroid tissue. Unfortunately, even with surgeons' abundant experience in thyroidectomies, unintentional injury or removal of PTGs is frequently identified due to the subjective and inconclusive localization of PTGs. Such accidental removal or injury of PTGs may lead to serious complications such as postoperative hypocalcemia or hypoparathyroidism. Therefore, there is a clear need to provide surgeons with intraoperative surgical guidance to safely identify PTGs in order to prevent the risk of surgical complications.

To meet this need, we aim to assess the ability of a new non-invasive, probe-based Hand-Held Imager (HHI) [hANDY-i, Optosurgical, LLC] to identify PTGs intraoperatively in order to help surgeons safely preserve PTGs in surgeries. Using Near-Infrared Autofluorescence Imaging (NIRAF), HHI's camera system will detect spontaneous autofluorescence signals without injection of any contrast. The probe component of the HHI will allow surgeons to conveniently and noninvasively navigate deeper areas where PTGs are difficult to reach. Should the HHI be able to discriminate PTGs from surrounding anatomical structures in the neck, the investigators hypothesize that surgeons will be better equipped to distinguish surgical margins of pathological tissue for safe resection in challenging thyroid surgeries.

Furthermore, in order to confirm the perfusion status of the PTGs indocyanine green (ICG) angiography imaging will be utilized in select cases where the blood supply deemed to be compromised, this will enable the surgeon to decide if the gland is still viable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thyroid tumors, or other conditions requiring thyroid surgery where frozen section biopsy of PTGs is deemed necessary under the surgeon's estimation.
* Plan for surgical resection of pathological PTGs.
* Subject age 18 - 70 yo.
* Subject agreement to participate

Exclusion Criteria:

* Not eligible for endocrine surgeries
* Plan for biopsy only of thyroid tumor (likely difficult to obtain sufficient tissue for both pathology analysis and study assessment)
* Subject age younger than 18 yo or older than 70 yo
* Subject refusal to participate
* Subject cognitively impaired and/or unable to provide assent.
* Allergy to indocyanine green and iodine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Number of Parathyroid Glands identified by the imager. | 10 minutes prior to injection of ICG
  Once the thyroid gland is removed the imager will be used to confirm the presence of 4 parathyroid glands, and will be compared to the number of parathyroid glands seen by naked eye.

SECONDARY OUTCOMES:
Perfusion assessment using ICG angiography. | 10 minutes after ICG injection.
  ICG angiography will be done for some of the patients, who have signs of perfusion insufficiency, 2 mg of ICG will be administered and glands will be observed by the imager to confirm if the blood flow is intact.
  Assessment will be measured as:
  0 - No signs of perfusion
  1. - Minimal perfusion
  2. - Well perfused
Measurement of Parathyroid hormone and calcium levels. | 1 day after the surgery.
  For all patients the levels of parathyroid hormone and calcium will measured pre and post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn Frazier, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data review for each subject will be completed shortly after enrollment. The research data will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by research staff will be secured and password protected. At the end of the study, all study databases will be archived at Johns Hopkins Hospital.

REFERENCES:
- [Result] Ali KM, Wolfe SA, Nagururu NV, Seo S, Han SM, Kim Y, Oh E, Kim DY, Ning B, Lee SY, Cha RJ, Tufano RP, Russell JO. Parathyroid gland detection using an intraoperative autofluorescence handheld imager - early feasibility study. Front Endocrinol (Lausanne). 2023 Jul 24;14:1190282. doi: 10.3389/fendo.2023.1190282. eCollection 2023. PMID 37554762
- [Result] Kim Y, Lee HC, Kim J, Oh E, Yoo J, Ning B, Lee SY, Ali KM, Tufano RP, Russell JO, Cha J. A coaxial excitation, dual-red-green-blue/near-infrared paired imaging system toward computer-aided detection of parathyroid glands in situ and ex vivo. J Biophotonics. 2022 Aug;15(8):e202200008. doi: 10.1002/jbio.202200008. Epub 2022 Apr 20. PMID 35340114

DOCUMENTS (1):
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT06939946/ICF_000.pdf